CLINICAL TRIAL: NCT02315469
Title: Pre-operative Assessment and Post-Operative Outcomes of Elderly Women With Gynecologic Cancers
Brief Title: Comprehensive Patient Questionnaires in Predicting Complications in Older Patients With Gynecologic Cancer Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NRG-CC002; NCI-2014-01376 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-ELD1301; NRG-CC002 (Other: NRG Oncology); NRG-CC002 (Other: DCP); NRG-CC002 (Other: CTEP); U10CA101165 (NIH); UG1CA189867 (NIH)
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Endometrial Serous Adenocarcinoma; Fallopian Tube Carcinoma; Malignant Female Reproductive System Neoplasm; Ovarian Carcinoma; Primary Peritoneal Carcinoma; Stage IIIA Uterine Corpus Cancer AJCC v7; Stage IIIB Uterine Corpus Cancer AJCC v7; Stage IIIC Uterine Corpus Cancer AJCC v7; Stage IVA Uterine Corpus Cancer AJCC v7; Stage IVB Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (geriatric assessment): At time of consent and within 14 days of surgery, patients complete a pre-operative geriatric assessment that evaluates functional status, comorbid medical conditions, psychological state, social support, and nutritional status. Post-operative complications are also collected for 6 weeks after surgery or until the date patients initiate or restart chemotherapy whichever is first.
  Interventions: Other: Comprehensive Geriatric Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Complete pre-operative geriatric assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies comprehensive patient questionnaires in predicting complications in older patients with gynecologic cancer undergoing surgery. Comprehensive patient questionnaires completed before surgery may help identify complications, such as the need for assistance in taking medications, decreased mobility, decreased social activity, and falls, and may improve outcomes for older patients with gynecologic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the preoperative geriatric assessment (GA)-gynecology (GYN) score will be associated with major post-operative complications in elderly patients undergoing open primary cytoreduction surgery.

SECONDARY OBJECTIVES:

I. To explore associations between individual variables of the preoperative geriatric assessment and major post-operative complications in patients undergoing open primary cytoreduction surgery.

II. To assess the association between the preoperative GA-GYN score and cytoreducibility defined by extent of residual disease in patients undergoing open primary cytoreduction surgery.

TERTIARY OBJECTIVES :

I. To evaluate whether the preoperative GA-GYN scores obtained before and after neoadjuvant chemotherapy will be associated with major postoperative complications in elderly patients undergoing open interval cytoreduction surgery.

II. To describe reasons why surgeons at centers where open cytoreduction surgery is the standard of care choose to perform interval surgery vs primary surgery, and to explore the association of the preoperative GA-GYN score with the decision to perform primary surgery or interval surgery or no surgery.

III. To collect the following specific information on how elderly women with suspected ovarian, fallopian tube, primary peritoneal carcinomas or advanced stage papillary serous uterine carcinoma are treated at centers that consider open cytoreduction surgery the standard of care: (1) the percentage of patients treated with primary open cytoreduction vs. interval open cytoreduction vs. no surgery and (2) to ascertain the extent of cytoreduction.

IV. To determine whether neoadjuvant chemotherapy will be associated with changes in the GA-GYN score to change by comparing the GA-GYN scores obtained before and after neoadjuvant chemotherapy.

V. To determine whether 30-day readmission rates after cytoreductive surgery correlate with the GA-GYN score.

OUTLINE:

At time of consent and within 14 days of surgery, patients complete a pre-operative geriatric assessment that evaluates functional status, comorbid medical conditions, psychological state, social support, and nutritional status. Post-operative complications are also collected for 6 weeks after surgery or until the date patients initiate or restart chemotherapy whichever is first.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected ovarian, fallopian tube, primary peritoneal carcinomas or advanced stage papillary serous uterine carcinoma irrespective of performance status; this clinical determination is made by the treating physician
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients who can understand sufficiently to be able to respond to questions posed by the study instruments
* Patients and/or caregiver (durable power of attorney) can give consent and caregiver can assist with the responses to questionnaire

  * NOTE: it is the intent of this trial that all patients 70 years or older presenting to the participating physician/center be offered enrollment onto this study; eligible patients may enroll and subsequently receive neoadjuvant chemotherapy followed by interval surgery, primary cytoreductive surgery or no surgery at all
* Post-operative pathology will not exclude patients from this study

Exclusion Criteria:

* Patients whose circumstances at the time of study entry do not permit completion of the study or required follow-up
* Patients who would have planned surgery performed by the minimally invasive technique; institutions which perform cytoreductive surgery via the minimally invasive technique should not participate in this study; the minimally invasive surgery (MIS) technique is also not considered standard technique for primary cytoreductive surgery for advanced stage ovarian, fallopian tube or peritoneal cancers
* Patients who receive chemotherapy treatment (for a gynecologic malignancy) prior to consideration of enrollment into this trial and taking the geriatric assessment will be excluded
* Patients who have a known pre-operative primary uterine cancer, confirmed by endometrial biopsy

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly women with suspected ovarian, fallopian tube, primary peritoneal or advanced stage papillary serous uterine carcinoma undergoing open cytoreductive surgery
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of major post-operative complications outlined in The American College of Surgeons' National Surgical Quality Improvement Program | Up to 6 weeks after surgery
GA-GYN score, defined as the summation of the risk score for each risk factor derived from the predictive model including 5 risk factors from the GA and 3 other risk factors | Up to 14 days before surgery
  Geriatric assessment variables are used in the predictive model; the risk factors will be used to derive the total score.

SECONDARY OUTCOMES:
Extent of residual disease in patients undergoing open primary cytoreduction surgery | 6 weeks after surgery
  The association between the preoperative GA-GYN score and cytoreducibility defined by extent of residual disease in patients undergoing open primary cytoreduction surgery will be assessed. Cytoreducibility is defined as complete cytoreduction (maximum dimension of residual disease =< 0.1 cm), optimal cytoreduction (maximum dimension of residual disease greater than 0.1 cm but less than or equal to 1.0 cm), or suboptimal cytoreduction (maximum dimension of residual disease greater than 1.0 cm) according to extent of residual disease.
Functional status, as measured by Instrumental Activities of Daily Living (IADL) | Up to 14 days before surgery
  The IADL subscale consists of 7 questions rated on a 3-point Likert scale measuring the degree to which an activity can be performed independently.
Functional status, as measured by Activities of Daily Living (ADL) | Up to 14 days before surgery
  The ALD uses a subscale of the Medical Outcomes Study physical health with 10 questions rated on a 3-point scale.
Patient's overall functioning, as measured by the physician rated performance rating scale | Up to 14 days before surgery
Patient's overall functioning, as measured by the self-reported performance rating scale | Up to 14 days before surgery
Number of falls in last 6 months | Up to 14 days before surgery
Comorbidity, as measured by the Older American Resources and Services (OARS) Physical Health section | Up to 14 days before surgery
  The OARS Physical Health Section is a comorbidity scale that contains a list of current illnesses and conditions an individual might have, and the degree to which they impair daily activities, rated on a 3-point scale of " not at all" to " a great deal."
Psychological status, as measured by the Mental Health Inventory (MHI) that is based upon the General Well-Being Scale | Up to 14 days before surgery
  The full length MHI consists of 38 items grouped into the following five subscales and three global scores: anxiety, depression, general positive affect, emotional ties, and loss of behavioral emotional control, Psychological Distress (negative affect), Psychological Well-Being (positive affect), and the MHI total score a 17 item version of the MHI will be used, which will yield three global scores of Psychological Distress, Psychological Well-Being and MHI total score, as in the original 38 item MHI.
Social functioning, as measured by the Medical Outcomes Study (MOS) Social Activity Limitations Measure | Up to 14 days before surgery
  The four-item subscale identifies the extent to which physical or emotional problems interfere with an individual's social activities. All items are rated on a 5-point Likert scale, with response categories varying in each item. The mean of the total score is transformed to a scale of 0-100, with a higher number indicating greater support.
Social support, as measured by the MOS Social Support Survey | Up to 14 days before surgery
Nutritional status, as measured by BMI | Up to 14 days before surgery
Nutritional status, as measured by percentage unintentional weight loss in last 6 months | Up to 14 days before surgery

OTHER OUTCOMES:
Frequency of reasons why surgeons perform interval surgery vs primary surgery and preoperative GA-GYN score | 6 weeks after surgery
Frequency of patients treated with primary cytoreduction, interval cytoreduction, no surgery and the extent of surgery | 6 weeks after surgery
Preoperative GA-GYN scores obtained before and after neoadjuvant chemotherapy | Up to 14 days before surgery
30-day readmission after cytoreduction surgery | Up to 30 days after surgery
  Will explore the correlation between pre-surgery GA-GYN score and dichotomized 30-day readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Amina Ahmed, Principal Investigator — NRG Oncology
Locations (393):
- United States (392):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Northside Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - Monongalia Hospital, Morgantown, West Virginia
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- McGill University Department of Oncology, Montreal, Quebec, Canada